CLINICAL TRIAL: NCT05822791
Title: Differences in ECG- vs. proLonged cardIac MonItor-DeTected Atrial Fibrillation in STROKE Patients
Brief Title: Differences in ECG- vs. proLonged cardIac MonItor-DeTected Atrial Fibrillation in STROKE Patients (DELIMIT AF-STROKE)
Status: Active, not recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: ReDA ID 13446
Record Dates: First submitted 2023-03-31; First posted 2023-04-21 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Atrial Fibrillation; TIA
MeSH Terms: conditions — Stroke; Atrial Fibrillation | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECG-Detected AF: Patients with atrial fibrillation detected on 12-lead ECGs done post-stroke
  Interventions: Diagnostic Test: ECG
- Device-Detected AF: Patients with atrial fibrillation detected on prolonged Holter monitoring lasting at least 7 days.
  Interventions: Diagnostic Test: Prolonged cardiac monitoring

INTERVENTIONS:
Diagnostic Test: Prolonged cardiac monitoring — Prolonged cardiac monitoring
  Groups: Device-Detected AF
Diagnostic Test: ECG — Electrocardiogram
  Groups: ECG-Detected AF

SUMMARY:
The present study is an investigator-initiated, single-center, retrospective study based on data from the London Ontario Stroke Registry (LOSR), aiming to compare the characteristics and outcomes of ECG-detected and Device-Detected atrial fibrillation in patients with ischemic stroke and transient ischemic attack.

DETAILED DESCRIPTION:
Patients with ischemic stroke and transient ischemic attack (TIA) without known atrial fibrillation (AF) are investigated with Prolonged Cardiac Monitoring (PCM) to detect AF. It is unclear if AF detected on 12-lead ECG after stroke occurrence bears the same risk of stroke as Device-detected AF. The investigators hypothesize, that Device-detected AF has a lower risk of ischemic stroke recurrence. The investigators will conduct a retrospective analysis of prospectively collected data from consecutive patients enrolled in the London Ontario Stroke Registry, (Ontario, Canada). The primary outcome will be a recurrent ischemic stroke at the end of the available follow-up window. The investigators will include ischemic stroke and TIA patients with ECG-detected AF and those with Device-detected AF on at least 7 days of Holter monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patient with a diagnosis of ischemic stroke or TIA.
* ECG-diagnosed AF or PCM-detected AF post ischemic stroke or TIA

Exclusion Criteria:

* Individuals younger than18 years-old
* Patients without IS or TIA diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an acute ischemic stroke or TIA in the London Ontario Stroke Registry without known AF, who are newly diagnosed with AF on a 12-lead ECG or a ≥7-day external cardiac monitor.
Sampling Method: Probability Sample
Enrollment: 366 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Recurrent Ischemic Stroke at End of available Follow-up Time | Duration of follow-up - minimum of 3 months after the first encounter with the stroke team
  Documented recurrent ischemic stroke

SECONDARY OUTCOMES:
Death | Duration of follow-up - minimum of 3 months after the first encounter with the stroke team
  Number of patients dead at the end of the available follow-up
Readmission for decompensated AF or heart failure | Duration of follow-up - minimum of 3 months after the first encounter with the stroke team
  Prevalence of readmission for decompensated AF or heart failure (HF) in each group
Prevalence of risk factors, cardiovascular comorbidities, and structural heart disease | Documented at baseline.
  Proportion with vascular risk factors, cardiovascular comorbidities, and structural heart disease in each group

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Sposato, MD, MBA (PI), Principal Investigator — London Health Sciences Centre, Western University (London, ON. Canada)
Locations (1):
- Heart & Brain Lab, Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual patients data will be made available upon reasonable request, conditional to approval from Western University Ethics Review Board